CLINICAL TRIAL: NCT04778059
Title: Phase 2 Trial to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Intravenous USB002 to Treat Patients With Respiratory Distress Due to COVID-19 Infection
Brief Title: Safety and Efficacy of USB002 for Respiratory Distress Due to COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll in timely manner due to nature of COVID
Sponsor: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USB002-2020-001
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: 2019 Novel Coronavirus Infection; COVID-19 Virus Infection; SARS Coronavirus 2 Infection; SARS-CoV-2 Infection; Respiratory Distress Syndrome, Adult; Adult Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- USB002 (Experimental)
  Interventions: Drug: USB002
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: USB002 — USB002 is pharmaceutically formulated Angiotensin 1-7 [A(1-7)], a non-hypertensive derivative of Angiotensin-II (A-II), and is suspended in a vehicle as a sterile solution of USB002. Depending upon cohort assignment, subjects in the USB002 group will receive one of four doses of USB002 administered intravenously (IV).
  Arms: USB002
Drug: Placebo — The placebo formulation will be the USB002 formulated solution without the addition of A(1-7). The placebo will be administered intravenously (IV).
  Arms: Placebo

SUMMARY:
This trial will study the use of USB002 given as an intravenous infusion in patients with respiratory distress due to infection with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from patient or legal representative;
2. Age 18 or greater;
3. Positive reverse transcription polymerase chain reaction (RT-PCR) for SARS-CoV-2 (≤10 days);
4. Respiratory rate > 20 RR;
5. SpO2 < 94% on room air, requiring supplemental oxygen, requiring invasive mechanical ventilation, or requiring ECMO;
6. Chest X-ray confirming bilateral pulmonary infiltrates;
7. Body mass index of ≤ 40 units/kg/m2;
8. Adequate method of birth control.

Exclusion Criteria:

1. Terminally ill patients due to underlying cardiac, cancer or severe debilitating neurological disease including coma;
2. Hospitalization expected to be < 96 hours due to medical improvement;
3. Interstitial lung disease;
4. Correction of QTc values obtained by 12 lead EKG using Fredericia's formula (QTcF) > 450 ms;
5. History of hypotension (mean arterial blood pressure < 65 mmHg), unrelated to CoVID-19 infection;
6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times upper limit of normal;
7. Participating concurrently on another clinical trial for the experimental treatment of COVID-19;
8. Active chemotherapy use;
9. Pregnant and/or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — The University of Arizona Health Sciences Center/ Banner Healthcare Systems Hospitals
Locations (1):
- The University of Arizona Health Sciences Center/ Banner Healthcare Systems Hospitals, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- USB002 90 ug/kg/Day: Subjects received standard of care plus a continuous IV infusion of 90 ug/kg/day USB002 for up to 96 hours.
- USB002 300 ug/kg/Day: Subjects received standard of care plus a continuous IV infusion of 300 ug/kg/day USB002 for up to 96 hours.
- USB002 600 ug/kg/Day: Subjects received standard of care plus a continuous IV infusion of 600 ug/kg/day USB002 for up to 96 hours.
- USB002 900 ug/kg/Day: Subjects received standard of care plus a continuous IV infusion of 900 ug/kg/day USB002 for up to 96 hours.
- Placebo: Subjects received standard of care plus a continuous IV infusion of USB002 placebo for up to 96 hours.
Period: Overall Study
Arm/Group | USB002 90 ug/kg/Day | USB002 300 ug/kg/Day | USB002 600 ug/kg/Day | USB002 900 ug/kg/Day | Placebo
Started | 3 | 3 | 3 | 2 | 10
Completed | 1 | 1 | 2 | 1 | 7
Not Completed | 2 | 2 | 1 | 1 | 3
Not completed — Death | 2 | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Telemed not done due to internal miscommunication. | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who received a USB002 or Placebo infusion were included in the analysis population for all outcomes analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | USB002 90 ug/kg/Day | USB002 300 ug/kg/Day | USB002 600 ug/kg/Day | USB002 900 ug/kg/Day | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (18.25) | 57.0 (8.66) | 61.0 (12.17) | 78.5 (0.71) | 59.8 (8.18) | 57.9 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 1 | 0 | 5
  Male | 1 | 3 | 1 | 1 | 10 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 0 | 5 | 10
  Not Hispanic or Latino | 1 | 2 | 1 | 2 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 2 | 2 | 10 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 2 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: Treatment emergent adverse events (including changes in laboratory assessments, physical examination findings, and vital signs)
Time Frame: Day 1 to Day 70 (or date of final measurement, if sooner)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | USB002 90 ug/kg/Day | USB002 300 ug/kg/Day | USB002 600 ug/kg/Day | USB002 900 ug/kg/Day | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 10
Participants | 2 | 3 | 2 | 2 | 8

ADVERSE EVENTS:
Time Frame: Up to 70 days
Description: AEs were collected at all study visits from the time of dosing.
Arm/Group | USB002 90 ug/kg/Day | USB002 300 ug/kg/Day | USB002 600 ug/kg/Day | USB002 900 ug/kg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 1/3 | 1/2 | 1/10
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 1/3 | 1/2 | 1/10
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 2/3 | 2/2 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | USB002 90 ug/kg/Day (N=3) | USB002 300 ug/kg/Day (N=3) | USB002 600 ug/kg/Day (N=3) | USB002 900 ug/kg/Day (N=2) | Placebo (N=10)
Withdrawal of life support (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Care Withdrawn
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Multiorgan dysfunction/Failure
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Brain Hemorrhage
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Worsening Covid Pneumonia
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Septic shock likely due to COVID-19 pneumonia and bacterial pneumonia
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Death, unknown
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Worsening hypotension secondary to septic shock
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Worsening hypercapnic respiratory failure requiring intubation and mechanical ventilation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | USB002 90 ug/kg/Day (N=3) | USB002 300 ug/kg/Day (N=3) | USB002 600 ug/kg/Day (N=3) | USB002 900 ug/kg/Day (N=2) | Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Per protocol, this clinical trial was designed to include two parts (Part 1 - dose escalation phase; Part 2 - dose expansion phase). Part 2 did not proceed due to enrolment difficulty. Sponsor encountered challenges in finding subjects that met study eligibility criteria. This was likely due to the role COVID-19 vaccinations played, limiting the spread and hospitalizations of COVID-19 patients. Sponsor terminated the trial early, when 21 subjects (all Part 1) had been enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT04778059/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT04778059/SAP_001.pdf